CLINICAL TRIAL: NCT04459338
Title: A Dose-response Study Examining the Contribution of GLP-1 Receptor Signaling to Glucagon-stimulated Insulin Secretion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adrian Vella (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Adrian Vella, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20-003995; 5R01DK126206-03 (NIH)
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Saline, Then Exendin-9,39 (Experimental): A week or two after screening, participants were admitted to the CRTU and Saline was infused during a hyperglycemic clamp during which escalating doses of glucagon were infused. After completion of this study participants underwent a washout period of 2 weeks after which they were readmitted to the CRTU and Exendin-9,39 was infused at 300pmol/kg/min was infused during a hyperglycemic clamp during which escalating doses of glucagon were infused.
  Interventions: Biological: Exendin-9,39; Other: Saline
- Exendin-9,39, Then Saline (Experimental): A week or two after screening, participants were admitted to the CRTU and Exendin-9,39 was infused at 300pmol/kg/min during a hyperglycemic clamp during which escalating doses of glucagon were infused. After completion of this study participants underwent a washout period of 2 weeks after which they were readmitted to the CRTU and Saline was infused during a hyperglycemic clamp during which escalating doses of glucagon were infused.
  Interventions: Biological: Exendin-9,39; Other: Saline

INTERVENTIONS:
Biological: Exendin-9,39 — Exendin-9,39 is a competitive antagonist of GLP-1 actions at the GLP-1 receptor
Other: Saline — Placebo comparator

SUMMARY:
The GLP-1 receptor (GLP1R) gene is found on the beta cells of the pancreas. Its role is in the control of blood sugar level by enhancing insulin secretion from the pancreas after eating a meal. The purpose of this research study is to evaluate the role of GLP1R in the response to elevated glucagon concentrations.

DETAILED DESCRIPTION:
Glucagon within the islet can signal the β-cell through GLP1R, and acts as an insulin secretagogue. This signaling is blocked by exendin-9,39. The relative importance of glucagon signaling through its cognate receptor or through GLP1R is unknown. Despite the lower affinity of GLP1R for glucagon, intra-islet concentrations of glucagon are sufficiently high to stimulate GLP1R. The other situation where this may occur is in response to pharmacologic doses of glucagon as used for β-cell function testing or raising peripheral glucagon concentrations above fasting values. The experiments proposed will characterize the role of GLP1R in glucagon's actions on the β-cell and the potential therapeutic role of dual (GLP-1R and glucagon receptor) agonists for the treatment of T2DM and obesity.

ELIGIBILITY:
Inclusion Criteria:

* 20 weight-stable, non-diabetic subjects

Exclusion Criteria:

* Age < 25 or > 65 years (to avoid studying subjects who could have latent type 1 diabetes, or the effects of age extremes in subjects with normal or impaired fasting glucose).
* HbA1c ≥5.9%
* Use of glucose-lowering agents.
* For female subjects: positive pregnancy test at the time of enrollment or study
* History of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
* Active systemic illness or malignancy.
* Symptomatic macrovascular or microvascular disease.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers responded to intramural advertising at the Mayo Clinic between March 2021 and September 2021
Pre-assignment Details: None of the enrolled subjects were excluded and all were randomized
Groups:
- Saline, Then Exendin-9,39: Subjects are admitted to the Clinical research unit the night before the study and the following morning after an overnight fast, at time 0 glucose is infused to raise concentrations to 165mg/dL. At the same time a glucagon infusion commences at 0.4ng/kg/min. At 60 min the infusion increases to 0.6ng/kg/min, at 120 min to 0.8ng/kg/min, at 180 min 1.0 ng/kg/min, and at 240 min 1.2 ng/kg/min. The glucagon infusion ends at 300 min. Saline infusion is started at time 0 and continues for 300 minutes.
  There is then a washout period of 14 days minimum
  Subjects are admitted to the Clinical research unit the night before the 2nd study and the following morning after an overnight fast, at time 0 glucose is infused to raise concentrations to 165mg/dL. At the same time a glucagon infusion commences at 0.4ng/kg/min. At 60 min the infusion increases to 0.6ng/kg/min, at 120 min to 0.8ng/kg/min, at 180 min 1.0 ng/kg/min, and at 240 min 1.2 ng/kg/min. The glucagon infusion ends at 300 min. Exendin-9,39 infusion is started at time 0 and continues for 300 minutes.
- Exendin-9,39, Then Saline: Subjects are admitted to the Clinical research unit the night before the study and the following morning after an overnight fast, at time 0 glucose is infused to raise concentrations to 165mg/dL. At the same time a glucagon infusion commences at 0.4ng/kg/min. At 60 min the infusion increases to 0.6ng/kg/min, at 120 min to 0.8ng/kg/min, at 180 min 1.0 ng/kg/min, and at 240 min 1.2 ng/kg/min. The glucagon infusion ends at 300 min. Exendin-9,39 infusion is started at time 0 and continues for 300 minutes.
  There is then a washout period of 14 days minimum
  Subjects are admitted to the Clinical research unit the night before the 2nd study and the following morning after an overnight fast, at time 0 glucose is infused to raise concentrations to 165mg/dL. At the same time a glucagon infusion commences at 0.4ng/kg/min. At 60 min the infusion increases to 0.6ng/kg/min, at 120 min to 0.8ng/kg/min, at 180 min 1.0 ng/kg/min, and at 240 min 1.2 ng/kg/min. The glucagon infusion ends at 300 min. Saline infusion is started at time 0 and continues for 300 minutes.
Period: Overall Study
Arm/Group | Saline, Then Exendin-9,39 | Exendin-9,39, Then Saline
Started | 5 | 6
Completed | 4 | 6
Not Completed | 1 | 0
Not completed — Loss of IV during study | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects without diabetes to enable evaluation of insulin secretory capacity
Groups:
- All Participants: All participants were randomized to receive all interventions
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Insulin Secretion Rate During Exendin-9,39 Infusion vs. Insulin Secretion Rate During Saline Infusion
Description: This is the area under the curve for insulin secretion over the duration of the hyperglycemic clamp (0 to 300 minutes during the study in the Clinical Research Unit).
Time Frame: Area under the curve was quantified at the end of the Saline Study and at the end of the Exendin-9,39 study
Measure: Mean (Standard Error); unit: nmol/min per 300 min
Groups:
- Insulin Secretion During the Saline Study: Subjects are admitted to the Clinical research unit the night before the study and the following morning after an overnight fast, at time 0 glucose is infused to raise concentrations to 165mg/dL. At the same time a glucagon infusion commences at 0.4ng/kg/min. At 60 min the infusion increases to 0.6ng/kg/min, at 120 min to 0.8ng/kg/min, at 180 min 1.0 ng/kg/min, and at 240 min 1.2 ng/kg/min. The glucagon infusion ends at 300 min. Saline infusion is started at time 0 and continues for 300 minutes.
- Insulin Secretion During the Exendin-9,39 Study: Subjects are admitted to the Clinical research unit the night before the study and the following morning after an overnight fast, at time 0 glucose is infused to raise concentrations to 165mg/dL. At the same time a glucagon infusion commences at 0.4ng/kg/min. At 60 min the infusion increases to 0.6ng/kg/min, at 120 min to 0.8ng/kg/min, at 180 min 1.0 ng/kg/min, and at 240 min 1.2 ng/kg/min. The glucagon infusion ends at 300 min. Exendin-9,39 infusion is started at time 0 and continues for 300 minutes.
Arm/Group | Insulin Secretion During the Saline Study | Insulin Secretion During the Exendin-9,39 Study
Number analyzed (Participants) | 11 | 10
nmol/min per 300 min | 191 (23) | 171 (19)
Statistical Analysis 1: Comparison: Insulin Secretion During the Saline Study vs Insulin Secretion During the Exendin-9,39 Study; All continuous data are summarized as means ± SEM. Area Under the Curve (AUC) was calculated using the trapezoidal rule. A paired, two-way Student t-test (parametric) or a Wilcoxon matched-pairs signed rank test (non-parametric) was used to examine differences between study days. A p-value <0.05 was considered statistically significant; Test type: Superiority; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Time between screening and completion of the study = 6 weeks
Groups:
- Saline: Subjects are admitted to the Clinical research unit the night before the study and the following morning after an overnight fast, at time 0 glucose is infused to raise concentrations to 165mg/dL. At the same time a glucagon infusion commences at 0.4ng/kg/min. At 60 min the infusion increases to 0.6ng/kg/min, at 120 min to 0.8ng/kg/min, at 180 min 1.0 ng/kg/min, and at 240 min 1.2 ng/kg/min. The glucagon infusion ends at 300 min. Saline infusion is started at time 0 and continues for 300 minutes.
- Exendin-9,39: Subjects are admitted to the Clinical research unit the night before the study and the following morning after an overnight fast, at time 0 glucose is infused to raise concentrations to 165mg/dL. At the same time a glucagon infusion commences at 0.4ng/kg/min. At 60 min the infusion increases to 0.6ng/kg/min, at 120 min to 0.8ng/kg/min, at 180 min 1.0 ng/kg/min, and at 240 min 1.2 ng/kg/min. The glucagon infusion ends at 300 min. Exendin-9,39 infusion is started at time 0 and continues for 300 minutes.
Arm/Group | Saline | Exendin-9,39
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 2/11 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline (N=11) | Exendin-9,39 (N=11)
Infusion line lost (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Phlebitis
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Nausea with glucagon infusion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT04459338/Prot_SAP_000.pdf